CLINICAL TRIAL: NCT05780008
Title: Eat My ABCs: Integrate Healthy Eating Into School Readiness
Brief Title: Eat My ABCs Project
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Michigan Health Endowment Fund (Other)
Responsible Party: Principal Investigator, Jiying Ling, Associate Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00008403
Record Dates: First submitted 2023-02-27; First posted 2023-03-22 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Nutrition, Healthy; Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This will be a one-group quasi-experimental design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eat My ABCs (Experimental): The experimental arm will receive the 14-week program including three main components: (1) "Eat My ABCs" child curriculum, (2) child fruit/vegetable letters to parents, and (3) program cookbook.
  Interventions: Behavioral: Eat My ABCs

INTERVENTIONS:
Behavioral: Eat My ABCs — The "Eat My ABCs" curriculum incorporates senses into learning (hear, see, smell, taste) and includes two sessions/week: 1) healthy eating learning; and 2) mindful food taste-testing activities to expose children to the one fruit, one vegetable, and relevant food items made from the one fruit and one vegetable to teach children the creative ways to make fruit/vegetable healthy and tasty.
  Child Letter to Parents. Every week, each child will create one letter, using stickers, regarding the one fruit and one vegetable presented in the program that he/she tasted or wanted to try at home.
  Program Cookbook. The investigators have developed a targeted program cookbook for low-income families. The program cookbook contains all budget-friendly recipes for healthy breakfasts, family meals, quick-fixes, kid-friendly snacks, and occasional sweets. In addition, the cookbook contains creative ways of making fruit/vegetable healthy, tasty, and kid-friendly at home.

SUMMARY:
Evaluate the effects of the "Eat My ABCs" program on improving Head Start preschoolers' eating behavior and anthropometric properties (BMI, percent body fat).

DETAILED DESCRIPTION:
The 14-week, community-led, program, aimed to establish lifelong healthy eating habits among vulnerable low-income preschoolers living in rural Michigan, includes three main components: (1) "Eat My ABCs" child curriculum, (2) child fruit/vegetable letters to parents, and (3) program cookbook.

"Eat My ABCs" Child Curriculum. Head Start teachers, along with teacher assistants/aids, will independently teach the age appropriate "Eat My ABCs" curriculum per week, for a total of 14 weeks. The "Eat My ABCs" curriculum follows the alphabet theme and incorporates the five senses into learning (hear fruit and vegetable information, see the color, feel the texture, smell the scent, and taste the flavor). Each week includes two sessions: 1) healthy eating learning on one fruit and one vegetable by incorporating school readiness knowledge on numbers, shapes, colors, and alphabets; and 2) food taste-testing activities to expose children to one fruit, one vegetable, and relevant food items made from the one fruit and one vegetable to teach children the creative ways to make fruit/vegetable healthy and tasty.

Child Letter to Parents. Every week, each child will create one letter, using stickers, regarding the one fruit and one vegetable presented in the program that he/she tasted or wanted to try at home.

Program Cookbook. The investigators have developed a targeted program cookbook for low-income families to overcome their limited cooking skills, busy schedules, and tight family budget. The program cookbook contains all budget-friendly recipes for healthy breakfasts, family meals, quick-fixes, kid-friendly snacks, and occasional sweets; and these recipes are culturally appropriate with a variety of choices such as American, Italian, Mexican, and Asian cuisines. In the cookbook, the investigators also promote slow /pressure-cooking recipes as using a slow or pressure cooker to prepare easy but healthy meals is an effective way to overcome low-income parent barriers of lack of time and cooking skills. In addition, the cookbook contains creative ways of making fruit/vegetable healthy, tasty, and kid-friendly at home.

ELIGIBILITY:
Inclusion Criteria:

* Any preschoolers aged 3-5 years old from the participating daycare classrooms.
* Having parental consent.

Exclusion Criteria:

* None

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Child's BMI | Change from week 0 (Time 1) to week 15 (Time 2)
  Height will be measured to the nearest 0.1cm using the Shorr board, and weight will be measured to the nearest 0.1kg using the Seca 874 scale or the BF-689 body fat/body water monitor. The online SAS program for Centers for Disease Control and Prevention Growth Charts was applied to calculate preschoolers' BMI for age and sex.
Percent body fat | Change from week 0 (Time 1) to week 15 (Time 2)
  Percent body fat will be measured to the nearest 0.1% using the BF-689 body fat/body water monitor. Each participant's biological sex, age, and height in cm were entered into the monitor for measuring % body fat. Trained data collectors then instructed participants to step onto the monitor surface and align feet with the four electrodes.
Skin carotenoids | Change from week 0 (Time 1) to week 15 (Time 2)
  An instrument called the Veggie Meter® will be utilized to assess skin carotenoids as an indicator for fruit/vegetable intake. To assess skin carotenoids in this study, each participant's non-dominant index finger will be used, and the average of three scans will be recorded as the final score.

SECONDARY OUTCOMES:
Parent fruit/vegetable/fiber intake | Change from week 0 (Time 1) to week 15 (Time 2)
  The 10-item Block Dietary Fruit/Vegetable/Fiber Screener will be used to assess parents' fruit/vegetable/fiber intake. A total score (range 0-50) will be calculated with a higher score indicating a higher intake of fruits and vegetables.
Household food insecurity | Change from week 0 (Time 1) to week 15 (Time 2)
  The U.S. Household Food Security Survey Module (19 questions) will be used. A total score (range 0-18) will be calculated with a higher score indicating a lower household food security.
Parental feeding skills | Change from week 0 (Time 1) to week 15 (Time 2)
  The Child Feeding Questionnaire (33 questions) will be used. Mean score (range 1-5) will be calculated for seven subscales including perceived responsibility for child feeding, perceived parent weight status, perceived child weight status, concerns about child weight, restriction of child's access to food, pressure to ask child to eat more food, and monitoring of child's eating. A higher mean score indicating a higher perceived feeding attitudes, beliefs, and practices.
Parental food resource management behavior | Change from week 0 (Time 1) to week 15 (Time 2)
  The 9-item Expanded Food and Nutrition Education Program Checklist will be used. A mean score (range 1-5) will be calculated with a higher mean score indicating a higher parental food resource management behavior.
Home eating environment | Change from week 0 (Time 1) to week 15 (Time 2)
  The 10-item Family Nutrition and Physical Activity Screening Tool will be used. A total score (range 10-40) will be calculated with a higher score indicating a healthier home eating environment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northeast Michigan Community Service Agency, Alpena, Michigan
  - Northwest Michigan Community Action Agency, Kalkaska, Michigan

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data can be shared with request.

REFERENCES:
- [Derived] Ling J, Kao TA, Yang X. Impact of food accessibility on eating and anthropometric outcomes among rural parent-child dyads: a secondary data analysis of a mindful eating intervention. BMJ Open. 2025 Dec 31;15(12):e108076. doi: 10.1136/bmjopen-2025-108076. PMID 41475815